CLINICAL TRIAL: NCT06904105
Title: A Phase 3 Clinical Study to Evaluate the Efficacy and Safety of HRS-7535 Tablets in Subjects With Overweight or Obesity
Brief Title: A Trial of HRS-7535 Tablets in Subjects With Overweight or Obesity
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-7535-303
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRS-7535 Group (Experimental)
  Interventions: Drug: HRS-7535 Tablets
- HRS-7535 Placebo Group (Placebo Comparator)
  Interventions: Drug: HRS-7535 Placebo Tablets

INTERVENTIONS:
Drug: HRS-7535 Tablets — HRS-7535 tablets.
  Arms: HRS-7535 Group
Drug: HRS-7535 Placebo Tablets — HRS-7535 placebo tablets.
  Arms: HRS-7535 Placebo Group

SUMMARY:
The study is being conducted to evaluate the efficacy and safety of HRS-7535 in subjects with overweight or obesity.

ELIGIBILITY:
Inclusion Criteria:

1. On the day of signing the informed consent form, the age should be between 18 and 75 years old.
2. At the screening period, the Body Mass Index (BMI) should meet the criteria of ≥ 28.0 kg/m², or ≥ 24.0 kg/m² with at least one weight-related comorbidity, such as hyperglycemia, hypertension, dyslipidemia, obstructive sleep apnea, or non-alcoholic fatty liver disease.
3. The participant should have controlled their diet and exercise for 3 months or more prior to screening and randomization, and the weight change in the past 3 months should not exceed 5%.
4. Before the trial, the participants must voluntarily sign the informed consent form, fully understand the trial content, procedures and potential adverse reactions, and have the ability and willingness to comply with the protocol requirements to complete this study.

Exclusion Criteria:

1. At the screening period, relevant laboratory test results are abnormal.
2. Electrocardiogram (ECG) results at the screening period show clinically significant abnormalities.
3. Uncontrolled severe hypertension at the screening period.
4. Presence of endocrine diseases that may significantly affect the body weight.
5. History of acute or chronic pancreatitis.
6. History of significant gastrointestinal diseases.
7. Severe infections, significant trauma, or major surgery within 30 days prior to screening, as judged by the investigator.
8. Use of medications or treatments that may cause significant weight gain or loss within 90 days prior to screening.
9. Known or suspected abuse of alcohol or narcotics.
10. Any condition deemed by the investigator to be unsuitable for participation in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 556 (Actual)
Dates: Start 2025-04-09 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
The percentage change in body weight relative to the baseline. | The 50th week after administration.
The proportion of participants with a body weight reduction of ≥ 5% relative to the baseline. | The 50th week after administration.

SECONDARY OUTCOMES:
The proportion of participants with a body weight reduction of ≥ 10% relative to the baseline. | The 50th week after administration.
Adverse events (AEs). | About 52 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided